CLINICAL TRIAL: NCT03437954
Title: Outcomes of Post-operative Diet in Children Following Tonsillectomy and Adenoidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Georgetown_Univeristy_MC
Record Dates: First submitted 2018-01-24; First posted 2018-02-19 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Chronic Tonsillitis; Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard soft diet (Other)
  Interventions: Other: Diet modification
- Non-restricted diet (Other)
  Interventions: Other: Diet modification

INTERVENTIONS:
Other: Diet modification — Patients will be randomized to follow the standard post-tonsillectomy diet at our institution, which consists of soft foods for ten days, or will be in the non-restricted diet group following surgery.

SUMMARY:
This research is being done because it is not known which dietary recommendations are best to help patients recover after a tonsillectomy and/or adenoidectomy. The purpose of this study is to determine how diet after tonsil/adenoid surgery affects bleeding, pain, and oral intake.

DETAILED DESCRIPTION:
Currently it is not known which dietary recommendations are best to help patients recover after a tonsillectomy and/or adenoidectomy. Traditional standard of care is to recommend that patients be restricted to a soft diet post-operatively. However, the investigators believe that there may be benefit in allowing patients to eat a restriction-free diet. In this study, the investigators will compare the current standard of care verse a non-restricted diet. The purpose of this study is to determine how diet after tonsil/adenoid surgery affects bleeding, pain, and oral intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients 3-12 years undergoing tonsillectomy and/or adenoidectomy.

Exclusion Criteria:

-

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding | From time of surgery through postoperative day 10.
  Blood tinged sputum or hemoptysis reported by patient or patient caregiver to on call resident or at post operative appointment; blood clot or bleeding from tonsil bed observed objectively on physical examination.

SECONDARY OUTCOMES:
Pain | From time of surgery through postoperative day 10.
  Patient or patient caregiver report of pain at each post operative day using a validated Wong Baker FACES pain scale.
Days missed from normal activity | From time of surgery through postoperative day 10.
  Patient or patient care giver reported number of days spent absent from normal activity as noted at post operative visit.

CONTACTS AND LOCATIONS:
Overall Officials: Earl Harley, MD, Study Director — MedStar Georgetown University Hospital
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States